CLINICAL TRIAL: NCT05632159
Title: Effect of Intraoperative Magnesium Sulphate on the Occurrence of Postoperative Delirium and Insomnia in Patients Undergoing Lumbar Fixation
Brief Title: Effect of Intraoperative Magnesium Sulphate on the Occurrence of Postoperative Delirium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mona Hussein, Associate professor of Neurology, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: FMBSUREC/090122022/Abd-Elsadek
Record Dates: First submitted 2022-11-19; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Patients Undergoing Lumbar Fixation

STUDY DESIGN:
Intervention Model Description: Evaluating the effect of intraoperative administration of Magnesium sulphate on the occurrence of post-operative delirium and insomnia in those patients.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional anaesthesia group (Placebo Comparator): Induction of anesthesia will be done by injecting fentanyl 2 μg/kg, propofol1.5-2.5 mg/kg and atracurium 0.5 mg/kg for muscle relaxation.
  Interventions: Drug: conventional anaesthesia
- Mg sulphate group (Active Comparator): Induction of anesthesia will be done by injecting fentanyl 2 μg/kg, propofol1.5-2.5 mg/kg and atracurium 0.5 mg/kg for muscle relaxation. With extra administration of intraoperative Magnesium sulphate 30 mg /kg as loading dose over 10 min then 10 mg /kg/ has maintenance dose
  Interventions: Drug: Mg sulphate

INTERVENTIONS:
Drug: Mg sulphate — Induction of anesthesia will be done by injecting fentanyl 2 μg/kg, propofol1.5-2.5 mg/kg and atracurium 0.5 mg/kg for muscle relaxation. With extra administration of intraoperative Magnesium sulphate 30 mg /kg as loading dose over 10 min then 10 mg /kg/ has maintenance dose
  Arms: Mg sulphate group
Drug: conventional anaesthesia — Induction of anesthesia will be done by injecting fentanyl 2 μg/kg, propofol1.5-2.5 mg/kg and atracurium 0.5 mg/kg for muscle relaxation.
  Arms: conventional anaesthesia group

SUMMARY:
Anaesthesia-related complications and mortality have been significantly reduced in the last years.(1) Nevertheless, anaesthesia-related side effects, such as post-operative delirium and sleep disturbances should not be underestimated. These side effects are economically challenging because they may lead to prolonged hospital stay and change in lifestyle condition. (2) After general anesthesia' sleep disturbances frequently occur. They are featured by insomnia' hyperinsomnia' narcolepsy' and changed sleep structure. (3.4) There are a lot of risk factors associated with post-operative sleep disturbance such as patient age, preoperative comorbidity, severity of surgical trauma, postoperative pain, postoperative complications and presence of pre-operative fatigue and depression. (5) Insomnia is one of the most prevalent health problems during pre-operative period and after post-operative recovery. It can lead to increase incidence of post-operative complications such as delayed recovery , anxiety and delirium (6).

Post-operative delirium is also one of the most common complications following anaesthesia with frequency estimates ranging from 10 to 50%. It is defined as delirium occurring 24 to 72 hours after surgery. (7) There are multiple risk factors for developing postoperative delirium including pre-existing dementia, old age, medical co-morbidities, and psycopathological symptoms. The recognition and treatment of Post-operative delirium is critically important because postoperative delirium is associated with poor outcomes including functional decline, dementia, cognitive impairment, increased hospital length of stay , increased mortality ( 11% increasing in the risk of death at 3 months and up to a 17% increased risk of death at 1 year. (8)

Animal studies have found that Magnesium can regulate melatonin production which is a hormone that guide body sleep wake cycle (9) . Magnesium is an essential cofactor for many enzymatic reactions' especially those that are involved in energy metabolism and neurotransmitter synthesis. It is a cofactor involved in more than 300 enzyme systems' regulates diverse biochemical reactions in the body (10.11) .

Magnesium supplements were used to improve insomnia symptom among older people in a double blinded placebo controlled clinical trial(12). Low dietary Magnesium intake was found to be significantly associated with depression which is a potential risk factor for insomnia(13). Also using Magnesium sulphate as an adjuvant has been associated with significantly less analgesic requirements and reducing postoperative pain which can improve quality of sleep and decrease insomnia symptoms.(14)

AIM OF THE STUDY The aim of this work is to identify the potential predictors of postoperative delirium and insomnia in patients undergoing lumbar fixation under general anesthesia, and to evaluate the effect of intraoperative administration of Magnesium sulphate on the occurrence of post-operative delirium and insomnia in those patients.

DETAILED DESCRIPTION:
Study design and Participants:

This prospective randomized controlled trial will be carried out on 80 patients indicated for lumbar fixation. The selected patients will be randomly assigned to one of the following two groups; the first group will receive conventional general anaesthesia only (40 participants) (conventional anaesthesia group), and the second group will receive conventional general anaesthesia with extra administration of intraoperative magnesium sulphate (40 participants) (Mg sulphate group). Randomization will be carried out using a closed opaque envelope technique. The patients will be recruited from the Neurosurgery, Beni-Suef University Hospital, in the period from November, 2021 to May 2022.

Inclusion criteria:

1. ASA I-II patients undergoing lumbar fixation.
2. Male and female patients with age range between 20-70 years.

Exclusion criteria:

1. Patients having gross hemodynamic or ventilatory fluctuations during the operation.
2. Patients who develop postoperative shock, major bleeding or complication.
3. Patients with a history of chronic pain that may interfere with sleep
4. Patients with sleep apnea syndrome.
5. Patient with a history of neurodegenerative disease, concomitant medical or metabolic illness known to affect sleep (e.g., thyroid, chest or cardiac disorders).
6. Patients with a history of psychiatric disorders .
7. Patients with a current history of illicit drug use.
8. Patients using hypnotic, anxiolytic, or antipsychotic drugs .
9. Allergy to any of the drugs that will be used in the study.
10. Pregnancy.

The included patients will be subjected to the following

1. History taking regarding: demographics, BMI, and co-morbidities
2. Assessment of depression using Beck Depression inventory (BDI) scale (15) . It will be done for all included patients one day before surgery. BDI is one of the most widely used instruments for measuring the severity of depression. It is consisted of twenty-one questions about how the subject has been feeling in the last week. Each question has a set of at least four possible answer choices, ranging in intensity from 0 to 3. A score 0-9 indicates minimal depression, a score 10-18 indicates mild depression, a score 19- 29 indicates moderate depression and a score 30-63: indicates severe depression.
3. Assessment of fatigue using a fatigue questionnaire. It will be done for all included patients one day before surgery. It is a14-item fatigue scale that assess physical and mental fatigue. Items 1-7 represent physical while items 8-11represent mental fatigue. Each item was scored using a bimodal response system; better than usual or no more than usual = zero, worse than usual or much worse than usual = one. The total score is the sum all items. Scores for physical and mental fatigue are the sum of the representative items for each section. (16) .
4. Assessment of insomnia using Insomnia severity index (ISI). It will be done for all included patients one day before and two weeks after surgery.

   ISI is a 7-item instrument measuring the individual's perception of insomnia symptoms over the previous two weeks. The evaluated dimensions are (severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28). (17)
5. Assessment of postoperative delirium using Memorial delirium assessment scale (MDAS). It will be done for all included patients between 24 hours and 48 hours after surgery. MDAS is structured as a 10-item, 4-point clinician-rated scale (possible range 0-30) designed to quantify the severity of delirium in medically ill patients. This instrument measures relative impairment in domains itemized as follows: 1, awareness; 2, orientation; 3, short-term memory; 4, digit span; 5, attention capacity; 6, organizational thinking; 7, perceptual disturbance; 8, delusions; 9, psychomotor activity; and 10, sleep-wake cycle. Items are rated on a 4point scale from 0 (none) to 3 (severe) depending on the level of impairment, rendering a maximum possible score of 30. A score of 13 has been recommended as a cut-off for establishing the diagnosis of delirium with a sensitivity of 70.59% and a specificity of 93.75% (18) .
6. Assessment of pain using Visual Analogue Scale (VAS). It will be done for all included patients at the night of the first day after 12 hours of the surgery. It is a continuous scale for describing pain severity or intensity. It consists of a horizontal line usually 10 centimeters in length. The ends of the line are defined as the extremes of pain; such as 'no pain at all' and 'worst imaginable pain'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain (19) .
7. Neurophysiological assessment. Electroencephalography (EEG) and Quantitative electroencephalography (QEEG) will be done for all included patients before, and between 24 hours and 48 hours after surgery.

   EEG and QEEG will be carried out in the Neuro Diagnostic & Research Center (NDRC), Beni-Suef University Hospital, using Nihon Kohden EEG Japan machine combined with Neuroguide QEEG software.

   EEG recording will be carried out for 20 minutes in a quiet room while the subject is relaxed with their eyes closed for 5 minutes and opened for 5 minutes to insure a high arousal level. The EEG scalp electrodes will be applied according to the international 10-20 system using an ear lobe electrode as a reference. The absolute power of 5 electrodes (CZ, T3, T4, T5, T6,) will be studied in the following frequency bands: delta (0.5-3Hz), theta (4-7 Hz) and also the absolute power of (O1, O2) will be studied in delta theta and alpha (8-12 Hz) bands.
8. Anaesthesia technique

   * A routine preoperative check-up will be performed for all selected patients including routine hematological and biochemical testing, in addition to electrocardiograms .
   * On arrival to the operating theatre, 18 G intravenous cannula will be inserted and IV crystalloid fluids will be infused, the monitor will be attached to the patients to take preoperative readings of HR , NIBP , SpO2.
   * The patients will be randomly divided to one of two groups:

Group 1:

* Induction of anesthesia will be done by injecting fentanyl 2 μg/kg, propofol1.5-2.5 mg/kg and atracurium 0.5 mg/kg for muscle relaxation. Laryngoscopy and endotracheal intubation will be performed using oral cuffed tube lubricated with lidocaine jelly 2 %.
* Maintainance of anesthesia will be done using sevoflurane 1.5-2 %, and Mixture of O2 and Air (70:30).

Group 2:

* Induction of anesthesia will be done by injecting fentanyl 2 μg/kg, propofol1.5-2.5 mg/kg and atracurium 0.5 mg/kg for muscle relaxation. Laryngoscopy and endotracheal intubation will be performed using oral cuffed tube lubricated with lidocaine jelly 2 %. With extra administration of intraoperative Magnesium sulphate 30 mg /kg as loading dose over 10 min then 10 mg /kg/ has maintenance dose (20).
* Maintenance of anesthesia will be done using sevoflorane1.5-2% and mixture of O2 and Air (70: 30) .

Ventilation in both groups will be controlled artificially to maintain an endtidal partial pressure of carbon dioxide of 35-45 mmHg.

At the end of surgery, neuromuscular blockade will be reversed with IV neostigmine 0.04mg/kg and atropine 0.02 mg/kg, the trachea will be extubated when the patient respond to commands, all patients will be transferred to PACU, where they receive oxygen via face mask 3-4 L/min and will be monitored.

The following parameters will be evaluated and recorded by senior anesthesiologist unaware of the study protocol:

1. Depth of anesthesia
2. Duration of anesthesia
3. Hemodynamics of the patients including BP and HR, SPO2, and End tidal CO2 will be continuously monitored and recorded every 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I-II patients undergoing lumbar fixation.
2. Male and female patients with age range between 20-70 years.

Exclusion Criteria:

1. Patients having gross hemodynamic or ventilatory fluctuations during the operation.
2. Patients who develop postoperative shock, major bleeding or complication.
3. Patients with a history of chronic pain that may interfere with sleep
4. Patients with sleep apnea syndrome.
5. Patient with a history of neurodegenerative disease, concomitant medical or metabolic illness known to affect sleep (e.g., thyroid, chest or cardiac disorders).
6. Patients with a history of psychiatric disorders .
7. Patients with a current history of illicit drug use.
8. Patients using hypnotic, anxiolytic, or antipsychotic drugs .
9. Allergy to any of the drugs that will be used in the study.
10. Pregnancy.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
Insomnia | 2 Weeks
  Assessment of insomnia using Insomnia severity index
Postoperative delirium using Memorial delirium assessment scale (MDAS). | 2 days
  Assessment of postoperative delirium using Memorial delirium assessment scale (MDAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No